CLINICAL TRIAL: NCT03516643
Title: Improving Myocardial Perfusion in Refractory Angina. Extracorporeal Shockwave Myocardial Revascularization in a Large Prospective Cohort
Brief Title: Extracorporeal Shockwave Myocardial Revascularization in Refractory Angina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Gianluca Alunni, MD, Cardiologist, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Angina Refractory; Angina Pectoris
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shockwave (Experimental): Extracorporeal Shockwave treatment on Ischemic Myocardium
  Interventions: Other: Extracorporeal Shockwave Myocardial Revascularization

INTERVENTIONS:
Other: Extracorporeal Shockwave Myocardial Revascularization — extracorporeal shockwave in ischemic area evaluated by SPECT
  Other Names: ESMR

SUMMARY:
This is a prospective cohort study to examine the efficacy of ESMR application in patients with refractory angina despite optimal medical therapy, not suitable for further PCI or CABG. Characteristics such as angina class scores (CCS class score), nitroglycerin consumption and hospitalization were compared at baseline and 1, 6 and 12 months after ESMR therapy. The effect on cardiac perfusion was assessed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* history of coronary artery disease;
* refractory angina pectoris, defined as the persistence of a angina pectoris (Canadian Cardiovascular Society class ≥ 2) for more than 3 months, despite the use of optimal medical therapy (which included β blockers, calcium channel blockers, long-acting nitrates, ivabradine, ranolazine and trimetazidine, up-titrated to the maximal tolerated dose) and coronary disease not amenable for further revascularization (as determined by an interventional cardiologist and cardiac surgeon);
* stable maximal medical therapy for at least 6 weeks;
* stress-induced ischemia at baseline SPECT;
* left ventricular ejection fraction higher than 40%;
* age higher than 18 years.

Exclusion Criteria:

* myocardial infarction or unstable angina in the previous 3 months,
* acute myocarditis, pericarditis, left ventricular thrombus, cardiac malignancies, chronic pulmonary disease (including emphysema and pulmonary fibrosis), endocarditis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Improvement of myocardial perfusion | 6months after ESMR
  Reduction in stress-induced ischemia at SPECT

SECONDARY OUTCOMES:
Reduction of symptoms | 1, 6, 12 months
  Improvement of CCS class
Reduction of symptoms | 1, 6, 12 months
  Improvement of NYHA class
Reduction of symptoms | 1, 6, 12 months
  Reduction of oral nitrates need

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Alunni, Principal Investigator — Città della Salute e della Scienza of Torino

IPD SHARING:
Plan to Share IPD: No